CLINICAL TRIAL: NCT01323283
Title: Intervention Study of the Ergogenic, Anti-inflammatory and Obesity Inhibitory Effects of Omega-3 Fatty Acids in 8 Year Old Children
Brief Title: Study of Omega-3 Fatty Acids Regarding Ergogenic, Anti-inflammatory and Obesity Inhibitory Effects in 8 Year Old Children
Acronym: STOPP-8 OM3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Midsona AB (Unknown); Forskningsrådet för arbetsliv och socialvetenskap, FAS (Unknown)
Responsible Party: Principal Investigator, Claude Marcus, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STOPP-8 OM3
Record Dates: First submitted 2011-03-24; First posted 2011-03-25 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Lifestyle-related Condition; Overweight and Obesity; Essential Fatty Acid Deficiency
Keywords: Omega-3; physical activity; children; obesity; sedentary; accelerometry; BMI; fatty acids; inflammatory markers; intervention; randomized; double blind
MeSH Terms: conditions — Mental Disorders; Overweight; Obesity; Motor Activity; Sedentary Behavior | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 supplementation (Active Comparator): 50 % of all included children will be randomized to this arm and administered capsules containing an omega-3 fatty acid composition.
  Interventions: Dietary Supplement: Omega-3
- Placebo (Placebo Comparator): 50 % of included children will be randomized to this arm and will be administered placebo capsules for the 15 week intervention.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 — This group will receive capsules containing omega-3, omega-6 and vitamin E. The dosage is six capsules per day containing a total of 558 mg of eico-pentaenoic acid (EPA), 174 mg of docosahexaeonic acid (DHA), 60 mg of gamma-linolenic acid (GLA) and 9,6 mg vitamin E in natural form (alfa-tocopherol), gelatine, glycerol. Participants will be instructed to eat three capsules each morning and evening.
  Other Names: OM3
  Arms: Omega-3 supplementation
Dietary Supplement: Placebo — This group will receive capsules containing rape seed oil. Participants will be instructed to eat three capsules each morning and evening.
  Arms: Placebo

SUMMARY:
This study hypothesizes that supplementation of omega-3 fatty acids (OM3) can increase physical activity, inhibit rapid gain in body weight and BMI in both sedentary and normally active 8 year old children. The purpose is secondarily to explore patterns of associations between OM3 supplementation, baseline and follow-up levels in all studied parameters. The study also aims to study if basal levels of OM3 are correlated with physical activity and to study if there is an association between basal levels of OM3 and the effect of OM3 supplementation on physical activity. To study if there is an effect of OM3 supplementation on triglyceride and LDL cholesterol levels and to study if there are more pronounced effects on children with higher levels. To study if OM3 supplementation, compared with placebo reduce weight increase among children at risk to become overweight. To study if there is an association between effects of OM3 on physical activity, weight and risk markers in blood. To study if there are any gender differences.

ELIGIBILITY:
Inclusion Criteria:

* Children in second grade of Swedish primary school willing to participate

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 423 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Total physical activity | 15 weeks
  The childrens' physical activity will be monitored during 7 consequtive days at 0 and 15 weeks with tri-axial accelerometer.
Body mass | 15 weeks
  The childrens' body mass will be measured with standardized scales at 0 and 15 weeks.

SECONDARY OUTCOMES:
BMI | 15 weeks
  The childrens' height will be measured using standardised stadiometer at 0 and 15 weeks. Along with the bosy mass data individual BMI (kilograms/meters squared) will be calculated for each time point.
Cardiovascular risk markers | 15 weeks
  Blood samples is collected from all participants at 0 and 15 weeks. This will not be decisive for inclusion in the study. Local anaesthesia will be used and the children can choose not to leave blood. Fasting blood samples will be analyzed for LDL-C, HDL-C, tot-C, TG, hsCRP, TNF-α, IL-6, IL-1, PAI-1, Glucose, Insulin, fatty acids and FTO-gene expression.
Childrens reported quality of life | 15 weeks
  A validated questionnaire for self-report of subjective perception of quality of life are filled out by each child at 0 and 15 weeks with assistance of an adult (parent or caregiver).
Perceived motor skill | 15 weeks
  A validated questionnaire for subjective self-report of motor skills are filled out by each child at 0 and 15 weeks with assistance of an adult (parent or caregiver).
Self reported physical activity | 15 weeks
  A validated questionnaire for subjective self-report of physical activity will be filled out by each child at 0 and 15 weeks with assistance by parent or caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Marcus, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Universitetssjukhuset, Huddinge, Södermanland County, Sweden